CLINICAL TRIAL: NCT01618370
Title: Radium-223 Dichloride (Alpharadin) in Castration-Resistant (Hormone-Refractory) Prostate Cancer Patients With Bone Metastases
Brief Title: Radium(223) Dichloride (Alpharadin) in Castration-Resistant (Hormone-Refractory) Prostate Cancer Patients With Bone Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16216; 2012-000075-16 (EudraCT Number)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Prostatic Neoplasms
Keywords: Radium 223; Alpharadin; Prostate Cancer; Bone metastases; Castrate resistant prostate cancer; Hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium-223 dichloride (Experimental)
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (BAY88-8223) — One injection to be administered every 4 weeks up to 6 injections. The dose per injection is 50 kBq/kg body weight.

SUMMARY:
This study is a prospective, interventional, open-label, multi-center early access program for the use of Ra-223 Cl2 in HRPC/CRPC (Hormone refractory prostate cancer / Castrate resistant prostate cancer) patients diagnosed with bone metastasis and to collect additional short and long term safety data on the product.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Histologically or cytologically confirmed prostate cancer
* Patients diagnosed with progressive bone predominant metastatic CRPC/HRPC (Hormone refractory prostate cancer / Castrate resistant prostate cancer) with at least 2 skeletal metastases on imaging with no lung, liver, and/or brain metastasis (lymph node only metastasis is allowed)
* Progressive disease is defined either by:

  * The appearance of new bone lesions. If progression is based on new lesion(s) on imaging only without an increase in prostate specific antigen (PSA), PSA values from 3 assessments within the last 6 months must be provided; OR
  * In the absence of new bone lesions by 2 subsequent increases in serum PSA over previous reference value, which should not be more than 6 months before screening, each measured at least 1 week apart with the last PSA ≥ 5 ng/mL. (The reference value time point 1, is defined as the last PSA measured before increases are documented, with subsequent values obtained a minimum of 1 week apart. If the PSA at time point 3 is greater than the PSA at time point 2, then eligibility has been met. If the PSA at time point 3 is not greater than the PSA at time point 2 but the PSA value at time point 4 and/or time point 5 is greater than the PSA at time point 2, the patient is eligible assuming that other criteria are met)
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 - 2
* Adequate hematological, liver, and renal function

  * Absolute neutrophil count (ANC) ≥ 1.5 x10^9/L
  * Platelet count ≥ 100 x10^9/L
  * Hemoglobin ≥ 10.0 g/dL (100 g/L; 6.2 mmol/L)
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin > 25 g/L

Exclusion Criteria:

* Treatment with an investigational drug within previous 4 weeks, or planned during the treatment period or follow-up
* Eligible for first course of docetaxel, i.e., patients who are fit enough, willing, and who are located where treatment with docetaxel is available
* Treatment with cytotoxic chemotherapy within previous 4 weeks, or failure to recover from AEs (adverse events) due to cytotoxic chemotherapy administered more than 4 weeks previous (however, ongoing neuropathy is permitted)
* Prior hemibody external radiotherapy is excluded. Patients who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count and platelets
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or radium-223 dichloride) for the treatment of bony metastases
* Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer)
* Visceral metastases as assessed by abdominal or pelvic computed tomography (CT) (or other imaging modality based on institutional standard of care)
* Presence of brain metastases
* Lymphadenopathy exceeding 6 cm in short-axis diameter
* Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis
* Imminent or history of spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Patients with history of spinal cord compression should have completely recovered.
* Any other serious illness or medical condition, such as but not limited to:

  * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2
  * Cardiac failure New York Heart Association (NYHA) III or IV
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
* Fecal incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2012-07-22 (Actual); Primary Completion 2014-08-13 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Acute safety, variables will be summarized using descriptive statistics based on adverse events collection | From baseline to 30 days post-treatment
  Safety variables to be analyzed during the treatment period include: ECOG PS, Skeletal-related events, Treatment emergent Grade 3-4 AEs, any grade of treatment-related AEs and SAEs, Safety laboratory tests including hematology and serum chemistry
Long-term safety, variables will be summarized using descriptive statistics based on adverse events collection | From 30 days post-treatment up to 3 years
  Safety variables to be analyzed during the follow-up period include: Skeletal-related events, Treatment related AEs and SAEs, Secondary malignancies

SECONDARY OUTCOMES:
Brief Pain Inventory, as assessed by BPI-SF questionnaire (Brief Pain Inventory-Short Form) | From baseline up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (183):
- Belgium (7):
  - Bruges
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Kortrijk
  - Leuven
  - Ottignies
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Brno
  - Ostrava
  - Plzen - Bory
  - Prague
- Denmark (3):
  - Copenhagen
  - Herlev
  - Odense
- Finland (5):
  - Helsinki
  - HUS
  - Kuopio
  - Seinäjoki
  - Tampere
- France (15):
  - Angers
  - Avignon
  - Caen
  - Clermont-Ferrand
  - Grenoble
  - La Roche-sur-Yon
  - Lille
  - Montpellier
  - Paris
  - Poitiers
  - Saint-Herblain
  - Suresnes
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (27):
  - Freiburg Im Breisgrau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Erlangen, Bavaria
  - München, Bavaria
  - Bremen, City state Bremen
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Braunschweig, Lower Saxony
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Rostock, Mecklenburg-Vorpommern
  - Aachen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Recklinghausen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Chemnitz, Saxony
  - Dresden, Saxony
  - Berlin, State of Berlin
  - Jena, Thuringia
  - Magdeburg
- Ireland (3):
  - Galway, Galway
  - Cork
  - Dublin
- Israel (9):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
  - Ẕerifin
- Italy (23):
  - Bari, Apulia
  - Brindisi, Apulia
  - Foggia, Apulia
  - Napoli, Campania
  - Forlì, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Pordenone, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Messina, Sicily
  - Trento, Trentino-Alto Adige
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Pisa, Tuscany
  - Padua, Veneto
  - Treviso, Veneto
  - Verona, Veneto
- Mexico City, Mexico City, Mexico
- Netherlands (5):
  - Alkmaar
  - Amsterdam
  - Leiden
  - Nijmegen
  - Zwolle
- Norway (5):
  - Ålesund
  - Bergen
  - Bodø
  - Lørenskog
  - Oslo
- Poland (2):
  - Bialystok
  - Warsaw
- Russia (2):
  - Moscow
  - Obninsk
- Spain (22):
  - A Coruña, A Coruña
  - Santiago de Compostela, A Coruña
  - Córdoba, Andalusia
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Santa Cruz de Tenerife, Canary Islands
  - Santander, Cantabria
  - Palma de Mallorca, Illes Baleares
  - Las Palmas de Gran Canaria, Las Palmas
  - León, León
  - Lugo, Lugo
  - Madrid, Madrid
  - Málaga, Málaga
  - Oviedo, Oviedo
  - Pamplona, Pamplona
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Valencia, Valencia
  - Madrid
  - Málaga
  - Zaragoza
- Sweden (10):
  - Eskilstuna
  - Kalmar
  - Karlstad
  - Linköping
  - Lund
  - Örebro
  - Stockholm
  - Sundsvall
  - Umeå
  - Uppsala
- Switzerland (8):
  - Aarau, Canton of Aargau
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Sankt Gallen, Canton of St. Gallen
  - Lausanne, Canton of Vaud
  - Zurich, Canton of Zurich
  - Bellinzona, Canton Ticino
  - Chur, Kanton Graubünden
- United Kingdom (27):
  - Bristol, Bristol
  - Cambridge, Cambridgeshire
  - Romford, Essex
  - Leicester, Leicestershire
  - Edinburgh, Lothian
  - Manchester, Manchester
  - Bebington, Merseyside
  - Northwood, Middlesex
  - Nottingham, Nottinghamshire
  - Taunton, Somerset
  - Sheffield, South Yorkshire
  - Guildford, Surrey
  - Sutton, Surrey
  - Coventry, Warwickshire
  - Birmingham, West Midlands
  - Wolverhampton, West Midlands
  - Aberdeen
  - Belfast
  - Cardiff
  - Derby
  - Glasgow
  - Hull
  - Leeds
  - London
  - Newcastle upon Tyne
  - Plymouth
  - Southampton

REFERENCES:
- [Derived] Saad F, Gillessen S, Heinrich D, Keizman D, O'Sullivan JM, Nilsson S, Miller K, Wirth M, Reeves J, Seger M, Carles J, Heidenreich A. Disease Characteristics and Completion of Treatment in Patients With Metastatic Castration-Resistant Prostate Cancer Treated With Radium-223 in an International Early Access Program. Clin Genitourin Cancer. 2019 Oct;17(5):348-355.e5. doi: 10.1016/j.clgc.2019.05.012. Epub 2019 May 31. PMID 31311763
- [Derived] Heidenreich A, Gillessen S, Heinrich D, Keizman D, O'Sullivan JM, Carles J, Wirth M, Miller K, Reeves J, Seger M, Nilsson S, Saad F. Radium-223 in asymptomatic patients with castration-resistant prostate cancer and bone metastases treated in an international early access program. BMC Cancer. 2019 Jan 7;19(1):12. doi: 10.1186/s12885-018-5203-y. PMID 30612558
- [Derived] Saad F, Carles J, Gillessen S, Heidenreich A, Heinrich D, Gratt J, Levy J, Miller K, Nilsson S, Petrenciuc O, Tucci M, Wirth M, Federhofer J, O'Sullivan JM; Radium-223 International Early Access Program Investigators. Radium-223 and concomitant therapies in patients with metastatic castration-resistant prostate cancer: an international, early access, open-label, single-arm phase 3b trial. Lancet Oncol. 2016 Sep;17(9):1306-16. doi: 10.1016/S1470-2045(16)30173-5. Epub 2016 Jul 26. PMID 27473888